CLINICAL TRIAL: NCT01564082
Title: Comparison of Early Endotracheal Tube Insertion With GlideScope Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Timothy Turkstra, Associate Professor and Staff Anesthesiologist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18855
Record Dates: First submitted 2012-03-06; First posted 2012-03-27 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Endotracheal Intubation
Keywords: endotracheal intubation; GlideScope

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ETT first (Experimental): Patients will have the endotracheal tube (ETT) introduced into the pharynx prior to GlideScope insertion, and then advanced under GlideScope guidance into the trachea.
  Interventions: Device: ETT First (GlideScope)
- Control Group (No Intervention): Patients will have the GlideScope introduced into the pharynx. The endotracheal tube (ETT) will then be advanced under direct vision into the mouth/pharynx. The ETT will then be advanced into the trachea under GlideScope guidance.

INTERVENTIONS:
Device: ETT First (GlideScope) — Patients will have the endotracheal tube (ETT) introduced into the pharynx under direct vision prior to GlideScope insertion. The ETT will then be advanced under GlideScope guidance into the trachea.
  Arms: ETT first

SUMMARY:
Patients presenting for elective surgery will be randomized to having the breathing tube inserted partly into the throat prior to GlideScope insertion, or having it inserted fully after GlideScope insertion.

DETAILED DESCRIPTION:
Patients presenting for elective surgery requiring orotracheal intubation will be randomized to having the Early Endotracheal Tube (ETT) inserted into the pharynx prior to GlideScope insertion and then having the ETT advanced under GlideScope guidance into the trachea, or, being intubated in the standard fashion with the GlideScope being inserted first and having the ETT then advanced via the pharynx into the trachea. The primary outcome is time to intubation.

ELIGIBILITY:
Inclusion Criteria:

1. Any adult patient booked for elective surgery requiring orotracheal intubation.
2. Any operator who has performed ≥ 20 GlideScope intubations.

Exclusion Criteria:

1. Any patient in whom the use of the GlideScope is contraindicated in the opinion of the attending anesthesiologist.
2. Any patient with cervical spine abnormalities.
3. Any patients with known or probable difficult airways.
4. Any patient requiring rapid sequence induction.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2012-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Time to Intubation | Day 1
  Duration of intubation of the patient

SECONDARY OUTCOMES:
Ease of intubation | Day 1
  Ease of intubation, measured on a Visual analog scale
Number of intubation attempts | Day 1
  Number of intubation attempts
Use of external laryngeal pressure | Day 1
  Use of external laryngeal pressure
Sore throat | Day 3
  Post operative sore throat, as rated by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy P Turkstra, MD, M. Eng., Principal Investigator — LHRI
Locations (2):
- Canada (2):
  - St. Joseph's Health Care, London, Ontario
  - London Health Sciences Center, London, Ontario